CLINICAL TRIAL: NCT03850392
Title: Effects of Local Cryotherapy on Cytokine, VRGF, NFkB and PG-E2 Levels in Knee Arthritis
Brief Title: Anti Inflammatory Effects of Local Cryotherapy in Knee Arthritis
Acronym: ALGGAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Xavier GUILLOT, Principal Investigator, Centre Hospitalier Universitaire de Besancon
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-A00848-35
Record Dates: First submitted 2019-02-18; First posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Arthritis Knee; Cryotherapy Effect
Keywords: cryotherapy; knee arthritis; cytokines
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: first phase : randomization ice versus cold CO2 second phase : ice-treated knees versus contralateral non-treated knees
Who Masked: Outcomes Assessor
Masking Description: the cytokine level assessment was blinded regarding the treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ice (Active Comparator): 16 knee arthritis patients treated by local ice (Thermogel®, Artsana, Grandate, Italy - 30 minutes application - twice within one single day).
  Just before the first cold application, at 9 a.m., and 24 hours later (day=1 at 9 a.m), an arthrocentesis was performed. Standard analyses were performed on the synovial fluid (bacteriology, cytology and microcrystal microscopic assessment). Furthermore, a part of the synovial fluid was centrifuged then frozen at -80°C. For the second arthrocentesis, after the synovial fluid was gathered for the same analyses, an intra-joint corticosteroid injection (Triamcinolone, HEXATRIONE®,Ethypharm, Saint-Cloud, France) was performed before removing the needle.
  Interventions: Device: cryotherapy (Thermogel - Artsana or Cryo+ - Cryonic)
- CO2 (Active Comparator): 16 knee arthritis patients treated by local hyperbaric cold CO2 at -78°C (Cryo+®, Cryonic, Salins-les-Bains, France - 2 minutes-applied twice within one single day). Just before the first cold application, at 9 a.m., and 24 hours later (day=1 at 9 a.m), an arthrocentesis was performed. Standard analyses were performed on the synovial fluid (bacteriology, cytology and microcrystal microscopic assessment). Furthermore, a part of the synovial fluid was centrifuged then frozen at -80°C. For the second arthrocentesis, after the synovial fluid was gathered for the same analyses, an intra-joint corticosteroid injection (Triamcinolone, HEXATRIONE®, Ethypharm, Saint-Cloud, France) was performed before removing the needle.
  Interventions: Device: cryotherapy (Thermogel - Artsana or Cryo+ - Cryonic)
- contralateral non-treated knees (No Intervention): 16 contralateral arthritic knees : the synovial fluid was collected and analysed according to the same procedure but no cold treatment was applied (while the corresponding contralateral arthritic knees were treated by ice) : At 9 a.m., and 24 hours later (day=1 at 9 a.m), an arthrocentesis was performed. Standard analyses were performed on the synovial fluid (bacteriology, cytology and microcrystal microscopic assessment). Furthermore, a part of the synovial fluid was centrifuged then frozen at -80°C. For the second arthrocentesis, after the synovial fluid was gathered for the same analyses, an intra-joint corticosteroid injection (Triamcinolone, HEXATRIONE®,Ethypharm, Saint-Cloud, France) was performed before removing the needle.

INTERVENTIONS:
Device: cryotherapy (Thermogel - Artsana or Cryo+ - Cryonic) — cold application (ice 30 min or cold CO2 2 min) twice during 1 day at an 8 hour-interval
  Arms: CO2; ice

SUMMARY:
47 patients with non-septic knee arthritis were treated by local ice (30 min) or cold CO2 (2 min) twice at an 8 hour-interval for 1 day.

The synovial fluid was collected just before the first cold application then 24 hours later.

Cytokine, VEGF, NF-kB, PG-E2 levels were assessed in the synovial fluid before/after treatment.

Contralateral arthritic knees were used as paired controls when possible.

DETAILED DESCRIPTION:
Patient inclusion Patients hospitalized in the rheumatology department in the Besançon university hospital in France and suffering from non-septic knee arthritis (rheumatoid arthritis according to the ACR-EULAR criteria, spondyloarthritis according to the ASAS criteria, gout or calcium pyrophosphate deposition disease (CPDD) - diagnosed by microscopic microcrystal assessment in synovial fluid) were included consecutively after signed informed consent. The protocol was declared and approved by the local ethic committee - clinicaltrials.gov:NCT02573298, Comité de Protection des Personnes - Est II: 12-664) and all research was performed in accordance with relevant guidelines/regulations. Patients suffering from septic arthritides and knee osteoarthritis were excluded. The patients had received no biologic treatment nor conventional DMARD for the 6 months preceding inclusion. Corticosteroids, colchicine and NSAIDs were stopped for at least 24 hours prior to inclusion.

Study design In the first phase of the study, the included patients were then randomized (1:1) to receive either local ice (Thermogel®, Artsana, Grandate, Italy - 30 minutes application - N=16) or hyperbaric cold CO2 at -78°C (Cryo+®, Cryonic, Salins-les-Bains, France - 2 minutes-N=16). Each patient received two applications of the randomly chosen technique at an 8 hour interval (9 a.m and 5 p.m). The skin temperature was monitored on the treated knee using MLT409/A Skin Temperature Probe® and ML309 Thermistor Pod® (ADInstruments,Dunedin, NZ). Thirty of these 32 patients were also included in another part of the study,aiming at evaluating the variations of the synovial power Doppler semi-quantitative score before/after 2 cold applications (ice versus cold CO2) 2. Just before the first cold application, at 9 a.m., and 24 hours later (day=1 at 9 a.m), an arthrocentesis was performed. Standard analyses were performed on the synovial fluid (bacteriology, cytology and microcrystal microscopic assessment). Furthermore, a part of the synovial fluid was centrifuged then frozen at -80°C. For the second arthrocentesis, after the synovial fluid was gathered for the same analyses, an intra-joint corticosteroid injection (Triamcinolone, HEXATRIONE®, Ethypharm, Saint-Cloud, France) was performed before removing the needle. These synovial fluid samples were used to perform the present part of the study, which was overall powered to evaluate the IL-6 level variations in the synovial fluid before/after 2 cold applications. After all the patients were included, synovial fluid IL-6, IL-17A, IL-1β, TNF-α, VEGF (Multiplex flow cytometry, CBA® BD Bioscience, Franklin Lakes, New Jersey, USA) and PG-E2 (ELISA, KGE004B®, Bio-Techne, Minneapolis, Minnesota, USA), NF-KB-P65/NFkB- p65-P (ELISA,85-86083-11®, Thermofisher, Waltham, Massachusetts, USA) levels were measured.

In the second phase of the study, we only included patients suffering from arthritides of both knees and treated them with local ice only, according to the protocol described above (N=15 +1 patient with knee bi-arthritis previously included in the first phase of the study in the ice treated group). The same protocol was applied to contralateral non-treated knees except cryotherapy treatment. Therefore, the synovial fluid was gathered and analyzed at the same evaluation times compared to treated knees, so these contralateral arthritic knees were used as paired controls for cytokine and enzyme assays (N=16).

Statistical analyses. The sample size was calculated in order to detect a significant variation in IL-6 synovialprotein levels before/after 2 cold applications. 15.78 (N=16) patients per group were necessary to detect a difference of 2325 pg/mL in IL-6 protein level with a power of 95% and a p-value of 0.05, according to published results of IL-6 assays in knee synovial fluid. Therefore, 2 groups of 16 patients were included in the first randomized phase of the study(ice versus cold CO2), then 16 patients with knee bi-arthritis were required for the second phase of the study (ice-treated versus contralateral knee, N=15+1 patient already enrolled in the first phase). For these reasons, a total of 47 patients were included. Paired Wilcoxon Mann-Whitney tests were performed in order to compare the mean cytokine and enzyme levels before/after treatment. Subgroup analyses were also planned (according to the treatment modalities (ice or cold CO2) and to the type of rheumatic disease (microcrystalinduced arthritides - pooled gout and CPDD patients - versus non-microcrystal-induced diseases - pooled RA and SpA patients). Furthermore, an interclass effect-size (weighted mean differences with 95% CI) for cytokine levels (before/after treatment) was calculated between ice-treated knees and the corresponding contralateral non-treated knees using R® software (rmeta® and meta® packages). Correlation tests were also performed using Pearson's coefficients in order to assess the parameters associated with cytokine level variations (before/after treatment). The statistical analyses were performed using R® and Graphpad® softwares.

Additional informations Funding: This work was supported by GIRCI Est II ("Young scientist" grant - 2014 - 21324 euros).

Competing interests: None.

ELIGIBILITY:
Inclusion Criteria:

* non-septic knee arthritis

Exclusion Criteria:

* biologic treatment within the last 6 months, septic arthritis

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-02-12 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
Il-6 protein level change in the synovial fluid (before / after treatment) | just before treatment (9 a.m) then 24 hours later (variation)
  Multiplex cytometry technique (pg/mL)

SECONDARY OUTCOMES:
pain Visual Analogic Scale change before / after treatment | just before treatment (9 a.m) then 24 hours later (variation)
  0 (minimum) -10 (maximum) numeric scale (0 : better - 10 : worse)
TNF-alpha change in the synovial fluid | just before treatment (9 a.m) then 24 hours later (variation)
  Multiplex cytometry (pg/mL)
IL-1 beta change in the synovial fluid | just before treatment (9 a.m) then 24 hours later (variation)
  Multiplex cytometry (pg/mL)
IL-17A change in the synovial fluid | just before treatment (9 a.m) then 24 hours later (variation)
  Multiplex cytometry (pg/mL)
VEGF change in the synovial fluid | just before treatment (9 a.m) then 24 hours later (variation)
  Multiplex cytometry (pg/mL)
NF-kB-p65 change in the synovial fluid | just before treatment (9 a.m) then 24 hours later (variation)
  ELISA (optical density)
phosphorylated NF-kB-p65 change in the synovial fluid | just before treatment (9 a.m) then 24 hours later (variation)
  ELISA (optical density)
PG-E2 change in the synovial fluid | just before treatment (9 a.m) then 24 hours later (variation)
  ELISA (optical density)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guillot X, Tordi N, Laheurte C, Pazart L, Prati C, Saas P, Wendling D. Local ice cryotherapy decreases synovial interleukin 6, interleukin 1beta, vascular endothelial growth factor, prostaglandin-E2, and nuclear factor kappa B p65 in human knee arthritis: a controlled study. Arthritis Res Ther. 2019 Jul 30;21(1):180. doi: 10.1186/s13075-019-1965-0. PMID 31362785